CLINICAL TRIAL: NCT06981624
Title: Comparaison d'un Traitement systématique à l'héparine Versus sélectif Pour la prévention de l'Occlusion Radiale EASY-Héparine
Brief Title: Comparison of the Systematic Versus the Selective Use of Heparin for the Prevention of Radial Artery Occlusion
Acronym: EASY-Heparin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Olivier F. Bertrand (Other)
Responsible Party: Sponsor-Investigator, Olivier F. Bertrand, MD, Laval University
Organization: Laval University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EASY-Heparin
Record Dates: First submitted 2025-05-01; First posted 2025-05-21 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-05

CONDITIONS: Radial Artery Occlusion
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heparin (No Intervention): Standard of care with 70-100 IU/kg of heparin after a diagnostic only trans-radial catheterization and a dual-artery compression device for hemostasis.
- No heparin (Experimental): No heparin administered after diagnostic only trans-radial catheterization and a dual-artery compression device for hemostasis.
  Interventions: Other: No heparin

INTERVENTIONS:
Other: No heparin — Hemostasis achieved using a dual-artery compression device without administration of heparin after trans-radial diagnostic catheterization
  Arms: No heparin

SUMMARY:
Randomized study comparing the systematic use of heparin (standard of care) against an elective use of heparin to prevent radial artery occlusion after a percutaneous catheterization using a dual-artery compression system.

ELIGIBILITY:
Inclusion Criteria:

* Any patient referred for a diagnostic transradial catheterism

Exclusion Criteria:

* Unable to understand study design or provide informed consent
* Unable to receive antiplatelet therapy with aspirina and/or clopidogrel-prasugrel and/or ticagrelor and intravenous anticoagulant derived from heparine or bivalirudine
* Local condition such as hematoma or pseudo-aneurims precluding radial or ulnar access.
* Presence of plethysmographic waveform with simultaneous radial and ulnar occlusive compression (due to colaterals or interouseous artery) precluding the evaluation of patent hemostasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rates of patent hemostasis | within 24 hours after diagnostic angiography
  Evaluation of patent hemostasis by pulse oximetry
Time to hemostasis | within 24 hours post-procedure
Nursing time involvement | within 24 hours post-procedure
  Calculation of nursing time required for surveillance and care of hemostasis
Evaluation of complications | within 30 days of procedure
  Compilation of access site complications such as radial artery occlusion, bleeding, presence and grading of hematomas, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- IUCPQ, Québec, Quebec, Canada